CLINICAL TRIAL: NCT06684808
Title: Impact of Active Breaks in the Classroom on Physical, Mathematical and Cognitive Performance in Elementary School Children
Brief Title: Impact of Active Breaks in Elementary School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Molise (Other)
Collaborators: Alessandra di Cagno (Unknown); Giuseppe Calcagno (Unknown); Giovanni Fiorilli (Unknown); Andrea Buonsenso (Unknown)
Responsible Party: Principal Investigator, Marco Centorbi, Principal Investigator, University of Molise
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 61/2020
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Physical Performance; Cognitive Performance; Academic Acheivement
Keywords: active breaks; children; academic achievement; physical activity; school time
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fitness (Experimental): The Fitness group engaged in active breaks aimed at improving cardiovascular efficiency. These breaks were designed to provide moderate to vigorous physical activity, incorporating both strength and aerobic exercises such as squats, jumping jacks, lunges, and running in place. Children were instructed to imitate the teacher's movements
  Interventions: Other: Fitness
- Creative (Experimental): The Creative group participated in active breaks that combined cognitive-creative and physical demands, incorporating activities like improvisations, dramatizations of events or short stories, simulation, and imitation games. These activities aimed to stimulate the creative process and enhance emotional expression within environmental constraints. Constraints, set by the teacher-such as specific rules, partner positioning, or speed of execution-limited movement options, encouraging students to explore new solutions to complete each task.
  Interventions: Other: Creative
- Combined (Experimental): The Combined group took active breaks by combining the Fitness protocol in the first break and the Creative protocol in the second.
  Interventions: Other: Combined
- Control (Active Comparator): Regular physical activity at school during the weeks.
  Interventions: Other: Control

INTERVENTIONS:
Other: Fitness — The Fitness group engaged in active breaks aimed at improving cardiovascular efficiency. These breaks were designed to provide moderate to vigorous physical activity, incorporating both strength and aerobic exercises such as squats, jumping jacks, lunges, and running in place. Children were instructed to imitate the teacher's movements.
  Arms: Fitness
Other: Creative — The Creative group participated in active breaks that combined cognitive-creative and physical demands, incorporating activities like improvisations, dramatizations of events or short stories, simulation, and imitation games. These activities aimed to stimulate the creative process and enhance emotional expression within environmental constraints. Constraints, set by the teacher-such as specific rules, partner positioning, or speed of execution-limited movement options, encouraging students to explore new solutions to complete each task.
  Arms: Creative
Other: Combined — The Combined group took active breaks by combining the Fitness protocol in the first break and the Creative protocol in the second.
  Arms: Combined
Other: Control — Regular physical activity at school during the weeks.
  Arms: Control

SUMMARY:
The purpose of the study was to evaluate the effects of 12 weeks of Active Breaks on motor, academic and cognitive performance in elementary school children.

DETAILED DESCRIPTION:
The purpose of the study was to evaluate the effects of 12 weeks of Active Breaks on motor, academic and cognitive performance in elementary school children. 159 children were recruited: 92 for experimental group (EG) and 67 for Control Group(CG); after the baseline assessment, the EG classes were randomly assigned into three experimental groups: creativity AB (CREAT; n = 30 ), fitness AB (FIT; n =31 ) and combined AB (COM; n= 31 ) . Specifically, the EG carried out an active break intervention for 12 weeks during curricular time, repeated twice a day, with the duration of 10 minutes, three times a week. CG did not performed any type of active breaks.

ELIGIBILITY:
Inclusion Criteria:

* attending second and third elementary classroom

Exclusion Criteria:

* to be free from injury, which could preclude the PA practice.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 159 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Height | after 12 weeks
Weight | after 12 weeks
Leaps forward on one foot | after 12 weeks
  Hopping forward on one foot along a line for 10 meters. This test consists of 4 items (what to do), each with specific execution criteria (what to observe). Generally, these criteria represent a mature execution pattern for that skill. Children receive 1 point if they perform the item correctly and 0 points if not
Side Gallop | after 12 weeks
  Gallop sideways for 10 meters. This test consists of 4 items (what to do), each with specific execution criteria (what to observe). Generally, these criteria represent a mature execution pattern for that skill. Children receive 1 point if they perform the item correctly and 0 points if not
Alternating forward hops on one foot | after 12 weeks
  Hopping forward by alternating the supporting foot for 10 meters. This test consists of 4 items (what to do), each with specific execution criteria (what to observe). Generally, these criteria represent a mature execution pattern for that skill. Children receive 1 point if they perform the item correctly and 0 points if not
Throwing a ball with one hand | after 12 weeks
  Throw the ball against the wall 10 meters away. This test consists of 4 items (what to do), each with specific execution criteria (what to observe). Generally, these criteria represent a mature execution pattern for that skill. Children receive 1 point if they perform the item correctly and 0 points if not
Receiving with the hands a thrown ball | after 12 weeks
  Catch the ball on the fly from a distance of 5 meters. This test consists of 4 items (what to do), each with specific execution criteria (what to observe). Generally, these criteria represent a mature execution pattern for that skill. Children receive 1 point if they perform the item correctly and 0 points if not
Hitting the ball with a tennis racket | after 12 weeks
  hitting the ball from a distance of 5 meters. This test consists of 4 items (what to do), each with specific execution criteria (what to observe). Generally, these criteria represent a mature execution pattern for that skill. Children receive 1 point if they perform the item correctly and 0 points if not
Long jump from a standing start | after 12 weeks
  Perform as long a forward jump as possible starting from a standing position.
Fast shuttle run 10x5m | after 12 weeks
  Run 5 m for 10 times at the highest possible speed
Assessment Test of Calculation Skills AC.MT 6-11 | after 12 weeks
  AC-MT 6-11 test proposes tests to ascertain the level of learning of calculus, basic assessment, and problem solving
Reynolds Interference Task (RIT) test | after 12 weeks
  Measurement of complex processing speed

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi del Molise, Campobasso, CB, Italy

IPD SHARING:
Plan to Share IPD: No